CLINICAL TRIAL: NCT04116463
Title: Testing the Effects of the CDSMP Among Lower-to-Middle Wage Workers
Acronym: SMARTLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0962; 1U48DP005017-01 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Chronic Disease
Keywords: lower-wage workers; chronic disease; self-management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Randomized at the individual level into intervention or attention-control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSMP (Experimental): Chronic Disease Self-Management Program (CDSMP) - a 6-week, group-based behavioral intervention delivered in a 2.5 hour session each week by a trained facilitator.
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP)
- Financial Self-Management (Active Comparator): Financial self-management course delivered in 3 modules, with a delivery time of approximately 1 hour per module.
  Interventions: Behavioral: Financial Self-Management Program (FSMP)

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Program (CDSMP)
  Other Names: Health Self-Management Program
  Arms: CDSMP
Behavioral: Financial Self-Management Program (FSMP)
  Arms: Financial Self-Management

SUMMARY:
The purpose of the proposed research is to extend the CDSMP to lower-wage populations aged 40-64 years by partnering with public libraries and employment support networks in select North Carolina counties. The specific aims of this research are to (1) test the effects of the CDSMP on employment and health outcomes among lower-wage working adults 40-64 years of age at 6 and 12 months from baseline, and explore the extent to which they are modified by select sociodemographic, chronic condition, and work-related factors, (2) conduct an economic evaluation of the CDSMP for employers (return on investment [ROI]), the health care system (ROI), and state governments (cost-effectiveness analysis (CEA)), and (3) assess factors associated with the reach, effectiveness, adoption, and implementation of the CDSMP among lower-wage workers using social marketing strategies designed to overcome program engagement and participation challenges that exist in this population.

DETAILED DESCRIPTION:
To evaluate the CDSMP's effect on key employment outcomes, an experienced team from the UNC-CH Prevention Research Center (PRC) will leverage its long-standing partnerships with employer networks, public libraries and community agencies throughout the state and the NC Division of Aging's network of 500 active CDSMP interventionists to conduct the proposed work. This research will produce new knowledge about CDSMP effects by (1) testing it in a high chronic disease burden population of employed, lower-wage adults in their preretirement years (ages 40-64), (2) focusing on employment productivity and cost-specific outcomes that would have direct relevance for employers, insurers, and policy-makers, and (3) targeting recruitment and CDSMP delivery to enhance uptake by lower-wage workers. The specific aims of the proposed study are to:

1. Test the effects of the CDSMP on employment and health outcomes among lower-wage working adults 40-64 years of age at 6 and 12 months from baseline, and explore the extent to which they are modified by select sociodemographic, chronic condition, and work-related factors. The primary study outcome is work productivity, measured as lost productivity time using Health and Work Performance Questionnaire (HPQ) absenteeism and presenteeism scores. Secondary study outcomes reflect health dimensions that are typically evaluated in relation to CDSMP delivery, and include measures of: chronic disease management self-efficacy, self management behaviors, health status, and healthcare utilization.
2. Conduct an economic evaluation of the CDSMP for employers (return on investment [ROI]), the health care system (ROI), and state governments (cost-effectiveness analysis [CEA]).
3. Assess factors associated with the reach, effectiveness, adoption, and implementation of the CDSMP among lower-wage workers using social marketing strategies designed to overcome program engagement and participation challenges that exist in this population.

ELIGIBILITY:
Inclusion Criteria:

* 40-64 years of age,
* residing within one of the 3 study counties,
* being employed 32 hours or more per week,
* being able to speak, read, and write in English,
* earning less than $60,000/year, and
* self-reporting having been diagnosed with at least one of the following chronic diseases: arthritis (osteoarthritis, rheumatoid, or gout); diabetes (Type I or II); cardiovascular disease; stroke; lung disease; chronic musculoskeletal-related pain; recurrent tension, migraine, or chronic daily headaches; HIV; Crohn's disease; depression; anxiety or panic attacks; post-traumatic stress disorder; or bipolar disorder.

Exclusion Criteria:

* unable to follow study instructions,
* severely disruptive, offensive, or socially inappropriate during group CDSMP workshops, or
* experiences an illness or injury during the study period that results in severe cognitive impairment.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Mean Work Limitations Questionnaire-25 Score 6M: Percent productivity loss due to presenteeism | 6 months
  The Work Limitations Questionnaire (WLQ) is a patient self-rated scale designed to assess on the- job impact of chronic health problems and/or treatment. The WLQ consists of 25 items in 4 dimensions: limitations handling time (5 items), physical work demands (6 items), mental interpersonal work demands (9 items), and output demands (5 items). Each item is rated on a 5- point scale from "All of the Time" (score 5) to "None of the Time" (score 0), or "Does Not Apply to My Job". The WLQ Productivity Loss Score is derived from the Global Productivity Index, which is calculated as a weighed sum of the 4 dimensions. Reduction in WLQ Productivity Loss score indicates less work limitation and represents the estimated percentage of productivity loss in the past two weeks due to presenteeism relative to a healthy benchmark sample. WLQ Productivity Loss Score ranges from 0% to 24.9%. Higher percent productivity loss reflects more severe work limitations.
Mean Work Limitations Questionnaire-25 Score 12M: Percent productivity loss due to presenteeism | 12 months
  The Work Limitations Questionnaire (WLQ) is a patient self-rated scale designed to assess on the-job impact of chronic health problems and/or treatment. The WLQ consists of 25 items in 4 dimensions: limitations handling time (5 items), physical work demands (6 items), mental interpersonal work demands (9 items), and output demands (5 items). Each item is rated on a 5- point scale from "All of the Time" (score 5) to "None of the Time" (score 0), or "Does Not Apply to My Job". The WLQ Productivity Loss Score is derived from the Global Productivity Index, which is calculated as a weighed sum of the 4 dimensions. Reduction in WLQ Productivity Loss score indicates less work limitation and represents the estimated percentage of productivity loss in the past two weeks due to presenteeism relative to a healthy benchmark sample. WLQ Productivity Loss Score ranges from 0% to 24.9%. Higher percent productivity loss reflects more severe work limitations.
Mean Work Limitations Questionnaire-4 Score 6M: Percent productivity loss due to absenteeism | 6 months
  The percentage of productivity lost due to work absences is the ratio of total missed work hours to total usual work hours in a two-week time frame. Both the numerator (total missed work hours due to health problems or medical care) and the denominator (total usual work hours) are computed based on information from four survey questions (two required and two optional), which are included in the WLQ Work Absence Module. Productivity loss due to absenteeism can range from 0% to 100%, with higher percent loss meaning more absenteeism.
Mean Work Limitations Questionnaire-4 Score 12M: Percent productivity loss due to absenteeism | 12 months
  The percentage of productivity lost due to work absences is the ratio of total missed work hours to total usual work hours in a two-week time frame. Both the numerator (total missed work hours due to health problems or medical care) and the denominator (total usual work hours) are computed based on information from four survey questions (two required and two optional), which are included in the WLQ Work Absence Module. Productivity loss due to absenteeism can range from 0% to 100%, with higher percent loss meaning more absenteeism.

SECONDARY OUTCOMES:
Mean Communication with Healthcare Provider Score 6M | 6 months
  3-item scale constructed by the CDSMP Stanford research team and used in the CDSMP National Evaluation (each item include 6-point Likert response scale (response range 0-5 per item)). Items reflect preparing list of questions to ask provider at visit, asking questions during the visit, discussing personal problems with provider during visits. Scores range from 0 to 15, with higher scores reflecting better communication.
Mean Communication with Healthcare Provider Score 12M | 12 months
  3-item scale constructed by the CDSMP Stanford research team and used in the CDSMP National Evaluation (each item include 6-point Likert response scale (response range 0-5 per item)). Items reflect preparing list of questions to ask provider at visit, asking questions during the visit, discussing personal problems with provider during visits. Scores range from 0 to 15, with higher scores reflecting better communication.
Medication adherence: Proportions and Means 6M | 6 months
  5 items internally constructed by research team members to reflect adherence over past month; proportions of participants in each group will be compared. Dichotomous items (No=0/Yes=1) include forgetting to take regularly scheduled medications, problems remembering to take regularly scheduled medication, stopping regularly scheduled medication when feeling better, stopping regularly scheduled medication when feeling worse. Participants responding they forgot to take regularly scheduled medication complete a 5th nominally-scaled item that asks how frequently they have forgotten to take in the past month (1 time =1, 2 times=2, 3 times=3, 4 times=4, 5 times=5, More than 5 times=6). Higher proportions on dichotomous items reflects worse within-group adherence. Higher mean scores on nominally-scaled item reflects worse within-group adherence.
Medication adherence Score: Proportions and Means 12M | 12 months
  5 items internally constructed by research team members to reflect adherence over past month; proportions of participants in each group will be compared. Dichotomous items (No=0/Yes=1) include forgetting to take regularly scheduled medications, problems remembering to take regularly scheduled medication, stopping regularly scheduled medication when feeling better, stopping regularly scheduled medication when feeling worse. Participants responding they forgot to take regularly scheduled medication complete a 5th nominally-scaled item that asks how frequently they have forgotten to take in the past month (1 time =1, 2 times=2, 3 times=3, 4 times=4, 5 times=5, More than 5 times=6). Higher proportions on dichotomous items reflects worse within-group adherence. Higher mean scores on nominally-scaled item reflects worse within-group adherence.
Mean Minutes per Week of Leisure Time Light or Moderate Exercise Score 6M | 6 months
  2 items that reflect the number of times per week engaged in light or moderate exercise during leisure time, and the number of minutes engaged in exercise for each occurrence; developed by CDSMP Stanford research team and used in CDSMP National Evaluation. Product of two items reflects total number of minutes per week, with possible ranges of 0 to 3360 (maximum score equivalent of 8 hours per day, 7 days per week). Higher scores = more favorable exercise profile.
Mean Minutes per Week of Leisure Time Light or Moderate Exercise Score 12M | 12 months
  2 items that reflect the number of times per week engaged in light or moderate exercise during leisure time, and the number of minutes engaged in exercise for each occurrence; developed by CDSMP Stanford research team and used in CDSMP National Evaluation. Product of two items reflects total number of minutes per week, with possible ranges of 0 to 3360 (maximum score equivalent of 8 hours per day, 7 days per week). Higher scores = more favorable exercise profile.
Mean Minutes per Week of Leisure Time Vigorous Exercise Score 6M | 6 months
  2 items that reflect the number of times per week engaged in vigorous exercise during leisure time, and the number of minutes engaged in exercise for each occurrence; developed by CDSMP Stanford research team and used in CDSMP National Evaluation. Product of two items reflects total number of minutes per week, with possible ranges of 0 to 3360 (maximum score equivalent of 8 hours per day, 7 days per week). Higher scores = more favorable exercise profile.
Mean Minutes per Week of Leisure Time Vigorous Exercise Score 12M | 12 months
  2 items that reflect the number of times per week engaged in vigorous exercise during leisure time, and the number of minutes engaged in exercise for each occurrence; developed by CDSMP Stanford research team and used in CDSMP National Evaluation. Product of two items reflects total number of minutes per week, with possible ranges of 0 to 3360 (maximum score equivalent of 8 hours per day, 7 days per week). Higher scores = more favorable exercise profile.
Mean Depressive Symptom Severity Score: Patient Health Questionnaire-8 6M | 6 months
  Valid and reliable instrument used in clinical settings to screen for possible depression. Includes 8 items, each with 4-point Likert responses that range from 0 to 3. Score range = 0 to 24, with higher scores reflecting more severe depressive symptoms.
Mean Depressive Symptom Severity Score: Patient Health Questionnaire-8 12M | 12 months
  Valid and reliable instrument used in clinical settings to screen for possible depression. Includes 8 items, each with 4-point Likert responses that range from 0 to 3. Score range = 0 to 24, with higher scores reflecting more severe depressive symptoms.
Mean Somatic Symptom Severity Score: Patient Health Questionnaire-15 6M | 6 months
  Valid and reliable instrument used in clinical settings to screen for somatization disorders. Includes 15 items, each with 3-point Likert responses that range from 0 to 2. Score range = 0 to 30, with higher scores reflecting more severe somatic symptoms.
Mean Somatic Symptom Severity Score: Patient Health Questionnaire-15 12M | 12 months
  Valid and reliable instrument used in clinical settings to screen for somatization disorders. Includes 15 items, each with 3-point Likert responses that range from 0 to 2. Score range = 0 to 30, with higher scores reflecting more severe somatic symptoms.
Mean Self-Rated Global Health Score: U.S. National Health Survey 6M | 6 months
  Single item of self-rated health with 5-point Likert response scale of 1 to 5. Higher score reflects poorer health rating.
Mean Self-Rated Global Health Score: U.S. National Health Survey 12M | 12 months
  Single item of self-rated health with 5-point Likert response scale of 1 to 5. Higher score reflects poorer health rating.
Mean Healthy Mental Health Days Score: Centers for Disease Control and Prevention 6M | 6 months
  Single item from BRFSS asking how many days out of past month mental health was not good. Possible range 0-31, with higher score reflecting worse mental health in past month.
Mean Healthy Mental Health Days Score: Centers for Disease Control and Prevention 12M | 12 months
  Single item from BRFSS asking how many days out of past month mental health was not good. Possible range 0-31, with higher score reflecting worse mental health in past month.
Mean Physical Health Days Score: Centers for Disease Control and Prevention 6M | 6 months
  Single item from BRFSS asking how many days out of past month physical health was not good. Possible range 0-31, with higher score reflecting worse mental health in past month.
Mean Physical Health Days Score: Centers for Disease Control and Prevention 12M | 12 months
  Single item from BRFSS asking how many days out of past month physical health was not good. Possible range 0-31, with higher score reflecting worse mental health in past month.
Mean Social Role Activity Limitation Score 6M | 6 months
  A 4-item scale developed by CDSMP research team at Stanford and used in CDSMP National Evaluation; each item with 5-point Likert response with item scores ranging from 0 to 4. Items reflect extent to which activities in the following social roles were limited due to health: activities with family / friends / neighbors / groups; hobbies or recreational activities; household chores; errands and shopping. Possible range of 0 to 16. Higher scores reflect more significant activity limitations due to health.
Mean Social Role Activity Limitation Score 12M | 12 months
  A 4-item scale developed by CDSMP research team at Stanford and used in CDSMP National Evaluation; each item with 5-point Likert response with item scores ranging from 0 to 4. Items reflect extent to which activities in the following social roles were limited due to health: activities with family / friends / neighbors / groups; hobbies or recreational activities; household chores; errands and shopping. Possible range of 0 to 16. Higher scores reflect more significant activity limitations due to health.
Mean Number of Times Hospitalized 6M | 6 months
  Single self-report item asking number of times hospitalized in past 3 months. Possible range 0 to 90. Higher score reflects greater hospitalization episodes.
Mean Number of Times Hospitalized 12M | 12 months
  Single self-report item asking number of times hospitalized in past 3 months. Possible range 0 to 90. Higher score reflects greater hospitalization episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn M Kneipp, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
UNC will prepare de-identified limited-access dataset suitable for sharing with other researchers. De-identification will include removal of obvious identifiers such as names and addresses. It will also include examination of less obvious potentially identifying variables. Continuous variables with extreme values may have the extremes truncated. Height and weight are examples of such variables. Categorical variables with small numbers of participants in some categories may have these categories pooled with larger categories.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available on December 31, 2019
Access Criteria: The limited-access dataset will be made available on the date specified. Data will be released as micro data. A researcher wishing to use the dataset will be required to obtain approval from UNC using an agreement form which clearly specifies the intended analyses as well as assurances that UNC policies and HIPPA regulations will be followed. If approval is granted, the dataset will be supplied on a CD, or whatever the most appropriate medium is at the time the dataset is prepared. The CD will contain the dataset in the form of .csv files. It will also include documentation describing the variables in the dataset and copies of the data collection forms used to collect the data.